CLINICAL TRIAL: NCT05917314
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effect of SlimBiotics Probiotic Formula on Weight Management and Metabolic Health Outcomes
Brief Title: A Study to Evaluate the Effect of SlimBiotics Probiotic Formula on Weight Management and Metabolic Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Slimbiotics (Unknown)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Organization: SlimBiotics Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 20317
Record Dates: First submitted 2023-06-01; First posted 2023-06-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Metabolic Health; Weight Loss; Stress; Well-Being, Psychological; Sleep; Healthy Eating
MeSH Terms: conditions — Weight Loss; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial. Participants will be randomized into the intervention group (SlimBiotics Probiotic) or into a placebo product control group.
Who Masked: Participant, Investigator
Masking Description: Both participant groups and the study coordinators will be blinded to the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (SlimBiotic Probiotic) (Experimental): Participants will take 1 serving (1 capsule) per day.
  Interventions: Other: Slimbiotic Probiotic
- Placebo Group (Placebo Comparator): Participants will take 1 serving (1 capsule) per day.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Slimbiotic Probiotic — SlimBiotics Probiotic formula contains three probiotic strains of L. fermentum:
  * Limosilactobacillus fermentum K7-Lb1
  * Limosilactobacillus fermentum K8-Lb1
  * Limosilactobacillus fermentum K11-Lb3 The product also contains Microcrystalline cellulose.
  Arms: Intervention Group (SlimBiotic Probiotic)
Other: Placebo — The placebo capsule contains microcrystalline cellulose.
  Arms: Placebo Group

SUMMARY:
This study is to evaluate the efficacy of a probiotic supplement on weight management and metabolic health. This study will be conducted as a hybrid trial consisting of both in-person visits and virtual assessments. Two groups will be included: the intervention (SlimBiotics Probiotic) and placebo.

The SlimBiotics probiotic formula is the first plant-based probiotic targeting weight management and metabolic health. Other competing probiotics are isolated from humans (feces) but the strains in SlimBiotics were isolated from a fermented plant (millet porridge cereal).

This product contains 3 probiotic strains:

Limosilactobacillus fermentum K7-Lb1 Limosilactobacillus fermentum K8-Lb1 Limosilactobacillus fermentum K11-Lb3

ELIGIBILITY:
Inclusion Criteria:

* Women & Men
* 18+
* BMI between 25-32
* Generally healthy - don't live with any uncontrolled chronic disease
* Own a sleep-tracking device (smart watch etc.)

Exclusion Criteria:

* Any pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders.
* Anyone with known severe allergic reactions.
* Women who are pregnant, breastfeeding or attempting to become pregnant
* Unwilling to follow the study protocol.
* Subjects currently enrolled in another clinical study
* Subjects having finished another clinical study within the last 4 weeks before inclusion
* Hypersensitivity, allergy or intolerance against any compound of the test products (e. g. acacia gum)
* Condition after implantation of a cardiac pacemaker or other active implants
* Sulfonylurea treatment
* Any disease or condition which might compromise significantly the hepatic (ascites), hematopoietic, renal, endocrine, pulmonary, central nervous, cardiovascular, immunological, dermatological, gastrointestinal or any other body system with the exception of the conditions defined by the inclusion criteria
* History of or present liver deficiency as defined by Quick < 70%
* Regular medical treatment including over-the-counter, which may have an impact on the study aims (e.g. probiotics containing supplements, laxatives, steroids etc.)
* History of hepatitis B, C, HIV
* Subjects who are scheduled to undergo any diagnostic intervention or hospitalization which may cause protocol deviations
* Simultaneous study participation by members of the same household
* Pregnancy and lactation
* Ascites as assessed by sonography
* Any diet to lose body weight
* Eating disorders or vegan diet
* Anorexia drugs
* Present drug abuse or alcoholism

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Visceral Fat Mass (VFM) [Time Frame: Baseline to Week 12] | 12 weeks
  VFM will be measured as an assessment of weight management.
Change in Body Weight [Time Frame: Baseline to Week 12] | 12 weeks
  Body weight will be measured as an assessment of weight management.
Change in Waist Circumference. [Time Frame: Baseline to Week 12] | 12 weeks
  Waist circumference will be measured as an assessment of weight management.
Change in blood pressure. [Time Frame: Baseline to Week 12] | 12 weeks
  Blood pressure will be measured as a marker of metabolic health. Both both systolic and diastolic blood pressure will be measured.
Change in resting heart rate. [Time Frame: Baseline to Week 12] | 12 weeks
  Resting heart rate will be measured as a marker of metabolic health.
Changes in metabolic health symptoms. [Time Frame: Baseline to Week 12] | 12 weeks
  Survey based assessment (0-5 scale) of changes in metabolic health symptoms.
Changes in total cholesterol [Time Frame: Baseline to Week 12] | 12 weeks
  Total cholesterol will be assessed as part of a lipid panel blood test.
Changes in blood levels of triglycerides. [Time Frame: Baseline to Week 12] | 12 weeks
  Triglycerides will be assessed as part of a lipid panel blood test.
Changes in blood levels of high-density lipoprotein. [Time Frame: Baseline to Week 12] | 12 weeks
  Blood levels of high-density lipoprotein will be assessed as part of a lipid panel blood test.
Changes in blood levels of low-density lipoprotein. [Time Frame: Baseline to Week 12] | 12 weeks
  Blood levels of low-density lipoprotein will be assessed as part of a lipid panel blood test.
Changes in blood glucose. [Time Frame: Baseline to Week 12] | 12 weeks
  Blood glucose levels will be assessed via blood test.
Changes in blood insulin levels. [Time Frame: Baseline to Week 12] | 12 weeks
  Blood insulin levels will be assessed via blood test.
Changes in hbA1c. [Time Frame: Baseline to Week 12] | 12 weeks
  hbA1c will be assessed via blood test.
Changes in hs-high-sensitivity C-reactive protein (hsCRP). [Time Frame: Baseline to Week 12] | 12 weeks
  hsCRP will be assessed via blood test.
Changes in alanine transaminase. [Time Frame: Baseline to Week 12] | 12 weeks
  Alanine transaminase will be assessed via blood test.
Changes in aspartate aminotransferase. [Time Frame: Baseline to Week 12] | 12 weeks
  Aspartate aminotransferase will be assessed via blood test.
Changes in gamma-glutamyl transferase (GGT). [Time Frame: Baseline to Week 12] | 12 weeks
  GGT will be assessed via blood test.

SECONDARY OUTCOMES:
Changes in sleep duration. [Time Frame: Baseline to Week 12] | 12 weeks
  Changes in sleep duration will be assessed by the participants using their own smart device (e.g. sleep tracker, Apple Watch, FitBit etc)
Changes in participants-perceived sleep quality. [Time Frame: Baseline to Week 12] | 12 weeks
  Changes in sleep quality will be assessed using study-specific surveys (0-5 scale).
Changes in participant-reported mental wellbeing. [Time Frame: Baseline to Week 12] | 12 weeks
  Mental well-being will be assessed study-specific surveys (0-5 scale).
Changes in scores on the Anxiety GAD7 Questionnaire [Time Frame: Baseline to Week 12] | 12 weeks
  Anxiety will be assessed using the validated Anxiety GAD7 Questionnaire (0-4 scale).
Changes in health eating habits. [Time Frame: Baseline to Week 12] | 12 weeks
  Changes in healthy eating habits and satiety will be assessed using the standardised Three-Factor Eating Questionnaire (0-4 scale).

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided